CLINICAL TRIAL: NCT04022720
Title: Role of Platelet-Rich Fibrin in Intraoral Soft Tissue Regeneration of Head and Neck Surgery Patients: A Prospective Clinical Trial
Brief Title: Platelet-Rich Fibrin in Intraoral Soft Tissue Regeneration
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled. Also, impacted of COVID on enrolling subjects hindered recruitment.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB201901614
Record Dates: First submitted 2019-07-12; First posted 2019-07-17 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: Mucosal Ulceration
Keywords: platelet rich fibrin (PRF)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet Rich Fibrin (PRF) Group (Experimental): Patients randomized to this group will receive treatment with a PRF graft.
  Interventions: Procedure: Platelet Rich Fibrin Application
- No Platelet Rich Fibrin Group (No Intervention): Participants in the observational control group will be managed at the time of the complication by standard of care methods.

INTERVENTIONS:
Procedure: Platelet Rich Fibrin Application — Platelet Rich Fibrin application at first post-op visit.
  Arms: Platelet Rich Fibrin (PRF) Group

SUMMARY:
Determine if the use of platelet rich fibrin (PRF) improves the rate and quality of healing for intraoral mucosal and epithelial soft tissue defects.

ELIGIBILITY:
Inclusion Criteria:

* Three categories of patients will be included in this study:

  1. Osteoradionecrosis (ORN) or medication related osteonecrosis of the jaw (MRONJ) patients who present to clinic with exposed bone and no clinical sign of infection.
  2. Patients having an excisional biopsy in clinic performed under local anesthesia resulting in a defect that cannot be easily repaired without compromising normal anatomy or function. These situations include excisions which would result in primary closure under tension or with distorted anatomy, require a local flap, or require healing by secondary intention.
  3. Patients presenting to the post-operative clinic with intraoral surgical wound dehiscence or an intraoral surgical wound healing by secondary intention.

     Exclusion Criteria:
* Patients under 18 years of age.
* Patient's unable to participate in blood draw either due to medical compromise, inability to tolerate the procedure, or inability of the physician to successfully draw the blood at the time of appointment.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-15 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Change in rate of healing in intraoral mucosa and epithelium soft tissues | 3 months post-operatively
  Improved healing times of PRF patients compared to control group.

CONTACTS AND LOCATIONS:
Overall Officials: Salam Salman, MD, DDS, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers